CLINICAL TRIAL: NCT02317900
Title: A Phase 1 Evaluation of the Safety and Protective Efficacy of a Single Dose of the Live Attenuated Tetravalent Dengue Vaccine TV005 to Protect Against Infection With Attenuated DENV-2, rDEN2∆30-7169
Brief Title: Evaluation of the Safety and Efficacy of a Single Dose of a Dengue Vaccine (TV005) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR 299
Record Dates: First submitted 2014-12-15; First posted 2014-12-17 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TV005 and rDEN2∆30-7169 (Experimental): Participants will receive one injection of TV005 at study entry (Day 0). On Day 180, participants will receive one injection of rDEN2∆30-7169.
  Interventions: Biological: TV005; Biological: rDEN2∆30-7169
- Placebo and rDEN2∆30-7169 (Placebo Comparator): Participants will receive one injection of placebo at study entry (Day 0). On Day 180, participants will receive one injection of rDEN2∆30-7169.
  Interventions: Biological: Placebo; Biological: rDEN2∆30-7169

INTERVENTIONS:
Biological: TV005 — TV005 is a live attenuated recombinant tetravalent dengue virus vaccine. It will be administered as a 0.5 mL dose containing 10^3 plaque forming units (PFUs) of each component (10^3.3 PFUs/mL of rDEN1∆30, 10^4.3 PFU/mL of rDEN2/4∆30(ME), 10^3.3 PFU/mL of rDEN3∆30/31-7164 and 10^3.3 PFU/mL of rDEN4∆30). It will be delivered by subcutaneous injection in the deltoid region of the upper arm.
  Arms: TV005 and rDEN2∆30-7169
Biological: Placebo — The placebo vaccine will be administered as a 0.5 mL dose delivered by subcutaneous injection in the deltoid region of the upper arm.
  Arms: Placebo and rDEN2∆30-7169
Biological: rDEN2∆30-7169 — rDEN2∆30-7169 is a live recombinant attenuated DENV-2 candidate vaccine virus. It will be administered as a 0.5 mL dose containing 10^3 PFUs of rDEN2∆30-7169. It will be delivered by subcutaneous injection in the deltoid region of the upper arm.

SUMMARY:
Dengue viruses are widespread in most tropical and subtropical regions of the world. This study will evaluate the safety and protective efficacy of a dengue vaccine (called TV005) against viremia and rash induced by a DENV-2 vaccine virus (called rDEN2∆30-7169) in healthy adults.

DETAILED DESCRIPTION:
There are four types of dengue viruses (DENV-1, DENV-2, DENV-3, and DENV-4), each of which can cause mild to life-threatening illness. This study will evaluate the protective efficacy of TV005 (a dengue virus vaccine) administered at Day 0 against viremia and rash induced by rDEN2∆30-7169 (a live attenuated candidate DENV-2 vaccine) administered at Day 180. The safety and immunogenicity of the TV005 and rDEN2∆30-7169 vaccines will also be evaluated.

This study will enroll healthy adults with no history of previous infection with a dengue virus or a flavivirus. Participants will be randomly assigned to receive a single injection of TV005 or placebo at study entry (Day 0). All participants will receive a single injection of rDEN2∆30-7169 on Day 180. For at least 30 minutes after each vaccination, participants will remain in the study clinic to be monitored for any adverse effects of the vaccines. Participants will record their temperature three times a day for 16 days after the first and second vaccinations.

In addition to study visits at Day 0 and 180, participants will attend study visits at Day 4, 6, 8, 10, 12, 14, 16, 21, 28, 56, 90, 150, 184, 186, 188, 190, 192, 194, 196, 201, 208, 236, 270, and 360. At select study visits, participants will undergo a physical examination, medical history review, blood collection, and a pregnancy test for female participants.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female between 18 and 50 years of age, inclusive
* Good general health as determined by physical examination, laboratory screening, and review of medical history
* Available for the duration of the study, approximately 26 weeks post-second inoculation
* Willingness to participate in the study as evidenced by signing the informed consent document
* Females Only: Female participants of childbearing potential willing to use effective contraception. Reliable methods of contraception include: hormonal birth control, condoms with spermicide, diaphragm with spermicide, surgical sterilization, intrauterine device, and abstinence (6 months or longer since last sexual encounter). All female participants will be considered having childbearing potential except for those with hysterectomy, tubal ligation, tubal coil (at least 3 months prior to vaccination), or post-menopausal status documented as at least 1 year since last menstrual period.

Exclusion Criteria:

* Females Only: Currently pregnant, as determined by positive beta-human choriogonadotropin (HCG) test, breastfeeding
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the requirements of the study protocol
* Screening laboratory values of Grade 1 or above for absolute neutrophil count (ANC), alanine aminotransferase (ALT), and serum creatinine, as defined in this protocol
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* Any significant alcohol or drug abuse in the past 12 months which has caused medical, occupational, or family problems, as indicated by participant history
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization within the last 6 months)
* HIV infection, by screening and confirmatory assays
* Hepatitis C virus (HCV) infection, by screening and confirmatory assays
* Hepatitis B virus (HBV) infection, by hepatitis B surface antigen (HBsAg) screening
* Any known immunodeficiency syndrome
* Use of anticoagulant medications
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 28 days prior to or following vaccination. Immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg prednisone equivalent per day for greater than or equal to 14 days.
* Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 28 days following vaccination
* Asplenia
* Receipt of blood products within the past 6 months, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 28 days following vaccination
* History or serologic evidence of previous dengue virus infection or other flavivirus infection (e.g., yellow fever virus, St. Louis encephalitis virus, West Nile virus)
* Previous receipt of a flavivirus vaccine (licensed or experimental)
* Anticipated receipt of any investigational agent in the 28 days before or after vaccination
* Participant has definite plans to travel to a dengue endemic area during the study
* Refusal to allow storage of specimens for future research

Inclusion Criteria for Second Vaccine:

* Good general health as determined by physical examination and review of medical history
* Available for the duration of the study, approximately 26 weeks after the second dose
* Willingness to participate in the study as evidenced by signing the informed consent document
* Females Only: Female participants of childbearing potential willing to use effective contraception for the duration of the trial. Reliable methods of contraception include: hormonal birth control, condoms with spermicide, diaphragm with spermicide, surgical sterilization, intrauterine device, and abstinence (6 months or longer since last sexual encounter). All female participants will be considered having childbearing potential except for those with hysterectomy, tubal ligation, tubal coil (at least 3 months prior to vaccination), or post-menopausal status documented as at least 1 year since last menstrual period.

Exclusion Criteria for Second Vaccine:

* Anaphylaxis or angioedema following the first dose of vaccine
* Females Only: Currently pregnant, as determined by positive beta-HCG test, breastfeeding
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the requirements of the study protocol
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* Any significant alcohol or drug abuse in the past 12 months which has caused medical, occupational, or family problems, as indicated by participant history
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization within the last 6 months)
* HIV infection, by screening and confirmatory assays
* HCV infection, by screening and confirmatory assays
* HBV infection, by HBsAg screening
* Any known immunodeficiency syndrome
* Use of anticoagulant medications
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 42 days prior to or following vaccination. Immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg prednisone equivalent per day for greater than or equal to 14 days.
* Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 28 days following vaccination
* Asplenia
* Receipt of blood products within the past 6 months, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 28 days following vaccination
* Anticipated receipt of any other investigational agent in the 28 days before or after vaccination
* Participant has definite plans to travel to a dengue endemic area during the study
* Refusal to allow storage of specimens for future research

Other Treatments and Ongoing Exclusion Criteria:

The following criteria will be reviewed on Study Days 28 and 56 following each vaccination. If any become applicable during the study, the participant will not be included in further immunogenicity evaluations, as of the exclusionary visit. The participant will, however, be encouraged to remain in the study for safety evaluations for the duration of the study.

* Use of any investigational drug or investigational vaccine other than the study vaccine during the 28-day period post-vaccination
* Chronic administration (greater than or equal to 14 days) of steroids (defined as prednisone equivalent of greater than to equal to 10 mg per day), immunosuppressants, or other immune-modifying drugs initiated during the 28-day period post-vaccination (topical and nasal steroids are allowed)
* Receipt of a licensed vaccine during the 28-day period post-vaccination
* Receipt of immunoglobulins and/or any blood products during the 28-day period post-vaccination
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Frequency of viremia in participants administered 10^3 PFU of rDEN2∆30-7169 at Study Day 180 | Measured through Day 360
  The incidence, magnitude, and duration of rDEN2∆30-7169 viremia following administration of rDEN2∆30-7169 at Study Day 180 in participants who received TV005 on Study Day 0 will be compared to those who received placebo on Study Day 0.
Proportion of participants who received TV005 & develop rash and/or neutropenia following administration of rDEN2∆30-7169 compared to proportion of participants who received placebo & developed rash and/or neutropenia following receipt of rDEN2∆30-7169 | Measured through Day 360

SECONDARY OUTCOMES:
Frequency of vaccine-related adverse events (AEs), graded by severity | Measured through Day 28 after each vaccination
  The frequency of immediate, systemic, and local AEs following vaccination will be summarized.
Frequency of virus-related AEs, graded by severity, following primary inoculation (inoculation of those participants who received placebo at Study Day 0) | Measured through Day 28 after each vaccination
  The frequency of immediate, systemic, and local AEs following vaccination of prior placebo-recipients with rDEN2∆30-7169 will be summarized.
Frequency of viremia of rDEN1∆30, rDEN2/4∆30(ME), rDEN3∆30/31, and rDEN4∆30 following TV005 vaccination | Measured through Day 16
  Quantity and duration of viremia will also be assessed
Number of TV005 vaccinees infected with DENV-1, DENV-2, DENV-3, and DENV-4 | Measured through Day 360
  Infection is defined as recovery of vaccine virus from the blood or serum of a participant and/or by seropositivity to DENV (PRNT50 greater than or equal to 1:10).
Evaluation of the immunogenicity of TV005, as assessed by PRNT50 to DENV-1, DENV-2, DENV-3, and DENV-4 at 28, 56, and 90 days after TV005 vaccination | Measured through Day 360
  Monovalent, bivalent, trivalent, and tetravalent seropositivity rates will be determined at these time points.
Evaluation of the immunogenicity of rDEN2∆30-7169 in flavivirus-naïve participants as assessed by the PRNT50 to DENV-2, for each participant at Study Day 0, 28, 56, and 90 post-vaccination with rDEN2∆30-7169 | Measured through Day 360
  This objective will be performed only for those participants who received placebo on Study Day 0 and rDEN2∆30-7169 on Study Day 180.
Number of rDEN2∆30-7169 vaccine recipients who become infected with DENV-2 following primary rDEN2∆30-7169 vaccination (placebo recipients at Study Day 0) | Measured through Day 360
  Infection is defined as recovery of vaccine virus from the blood or serum of a participant and/or by seropositivity to DENV-2 (PRNT50 greater than or equal to 1:10)
Evaluation of if peak neutralizing antibody titer against DENV-2 following TV005 vaccination or neutralizing antibody titer against DENV-2 measured at Day 180 correlates with protection against viremia, rash, and/or neutropenia following inoculation | Measured through Day 360
Evaluation of if inoculation with rDEN2∆30-7169 at 6 months will boost neutralizing antibody titers to DENV-1, DENV-2, DENV-3, and DENV-4 in those participants who received TV005 on Study Day 0. | Measured through Day 360

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research (CIR), Johns Hopkins School of Public Health
Locations (2):
- United States (2):
  - Center for Immunization Research, Johns Hopkins School of Public Health, Baltimore, Maryland
  - University of Vermont Vaccine Testing Center, Burlington, Vermont

REFERENCES:
- [Derived] Pierce KK, Durbin AP, Walsh MR, Carmolli M, Sabundayo BP, Dickson DM, Diehl SA, Whitehead SS, Kirkpatrick BD. TV005 dengue vaccine protects against dengue serotypes 2 and 3 in two controlled human infection studies. J Clin Invest. 2024 Feb 1;134(3):e173328. doi: 10.1172/JCI173328. PMID 37971871